CLINICAL TRIAL: NCT06221475
Title: A Two-part, Single Center, Open-label Study to Investigate the Pharmacokinetics, Metabolic Disposition, Mass Balance and Absolute Bioavailability of BAY 2927088 in Healthy Male Participants
Brief Title: A Study to Learn How BAY2927088 is Taken up and Handled by the Body in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22249; 2022-502771-38-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-05

CONDITIONS: Advanced Non-small Cell Lung Cancer; EGFR Mutation; HER2 Mutation; Healthy Volunteers
Keywords: NSCLC; TKI

STUDY DESIGN:
Intervention Model Description: This is a single-arm open-label, single dose study in healthy male participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy male participants from Netherlands (Experimental): In Part 1, participants will receive a single dose of 40 mg of BAY2927088 as oral tablets on Study Day 1 approximately 30 min after a light meal, they will then receive a single dose of a microtracer not exceeding 100 ug of [14C]-BAY2927088 and 37 kilo becquerel (kBq) [1000 nano Curie (nCi)] of 14C will be administered intravenously (IV) as a 15 min infusion ending at the expected median time to maximum concentration (tmax) for the tablet (2 hours oral post-dose). After 2 days of washout, participants will move on to Part 2. In Part 2, on Study Day 1 approximately 30 min after a light meal, all enrolled participants will receive a single dose of 40 mg BAY2927088 containing approximately 3.7 MBq (100 µCi) [14C]-BAY 2927088 administered as an oral solution
  Interventions: Drug: BAY2927088 coated tablet 10 mg; Drug: [14C]-BAY2927088 solution for infusion; Drug: [14C]-BAY2927088 oral solution

INTERVENTIONS:
Drug: BAY2927088 coated tablet 10 mg — 4 coated tablets (10 mg) per single dose 30 min after a light meal
Drug: [14C]-BAY2927088 solution for infusion — IV infusion 15 min ending at 2 hours oral post-dose
Drug: [14C]-BAY2927088 oral solution — After a light meal

SUMMARY:
Researchers are looking for a better way to treat men who have advanced non-small cell lung cancer (NSCLC). NSCLC is a group of lung cancers that have spread to nearby tissues or to other parts of the body.

Epidermal growth factor receptor (EGFR) and human epidermal growth factor receptor 2 (HER2) are proteins that help cells to grow and divide. A damage (also called mutation) to the building plans (genes) for these proteins in cancer cells leads to a production of abnormal EGFR and/or HER2. These abnormal proteins drive the growth and the spread of the cancer. Several EGFR and/or HER2 mutations exist in the cancer cells. The study treatment works by blocking the mutated EGFR and HER2 protein present in NSCLC cells and may help stop the further spread of NSCLC.

BAY2927088 is under development, once it is approved, it may help treat people with NSCLC.

The participants of this study will be healthy men and will have no benefit from the administration of BAY2927088. However, the study will provide important information for the design of subsequent studies with BAY2927088 in people with NSCLC.

The participants in this study will get the non-radiolabeled and radio-labeled study treatment BAY2927088 in the form of tablets and solution by mouth and as an intravenous infusion in the arm. By radiolabeling the study treatment, researchers can track its movement and breakdown in the body of the participants. During the study, the study team will do physical examinations, take medical history, ask the participants questions about their smoking or alcohol consumption habits and other medications used, check vital signs such as blood pressure, heart rate, body temperature and the number of breaths taken per minute (respiratory rate), take blood and urine samples, do HIV (human immunodeficiency virus), hepatitis and optional COVID-19 tests per local regulations, and examine heart health using electrocardiogram (ECG).

Each study participant will go through a first test phase (screening) of up to 28 days before the start of treatment. The study will have two parts. In part 1, the study participants will take a single dose of the non-radiolabeled study treatment in the form of tablets by mouth 30 minutes following a light meal. They will then receive the radiolabeled study treatment as an intravenous infusion in the arm over 15 minutes. After 2 days of washout, the same group of participants will move on to Part 2 of the study. They will take a single dose of the radio-labeled study treatment as a solution by mouth 30 minutes after a light meal. The participants and the study team know what treatment the participants will take. The total duration of the study will be approximately 8 weeks per participant, including an in house stay of approximately 23 days and 22 nights. There will be a final examination on the last day of their in-house stay before the participants are discharged and go home.

The study doctors and their team will contact the participant to learn about the participant's health until the participant completes the study.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Participant must be 18 or age of legal maturity to 55 years of age inclusive, at the time of signing the informed consent
* Participants who are overtly healthy as determined by the investigator or medically qualified designee based on medical evaluation including medical history, laboratory tests, physical, cardiac, and neurologic examination
* Body mass index (BMI) within the range [18 - 30] kg/m^2 (inclusive), with bodyweight above/equal to 50 kg
* Male
* Study participants of reproductive potential must agree to use adequate contraception when sexually active during the study period and for at least 3 months after the last dose of study intervention, and refrain from donating sperm during this period
* Participant must have venous access sufficient to allow blood sampling as required by the protocol
* Participant must be willing to undergo multiple blood draws as required by the protocol
* Participant must be willing to comply with dietary and fluid requirements during the treatment period (including abstaining from alcohol use)
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Existing relevant diseases of vital organs (e.g., liver diseases, heart diseases, gastrointestinal diseases, interstitial lung disease), central nervous system (for example seizures) or other organs (e.g., diabetes mellitus)
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study intervention will not be normal
* Any relevant diseases within 4 weeks prior to the first study intervention administration as judged by the investigator
* A medical history of risk factors for Torsades de pointes (e.g., family history of long QT syndrome) or other clinically significant arrhythmias as judged by the investigator
* Known history of hypersensitivity (or known allergic reaction) to BAY2927088-related compounds, or any components of the formulation
* History of known or suspected malignant tumors
* Participants with any type of psychiatric disorder, especially any mood disorders including medical history with suicidal ideation and/or suicide attempts, which may disable the participant to consent
* Any condition which may result in longer than usual retention of urine or feces in the body, such as pronounced (less than one defecation in 3 days) constipation or symptomatic prostatic hypertrophy
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton [excluding spinal column]), during work or during participation in a clinical study in the period of 1 year prior to screening
* Participant will be excluded when he participated in another study with a radiation burden of 0.1 - 1 mSv (inclusive) in the period of 1 year prior to screening; 1.1 - 2 mSv (inclusive) in the period of 2 years prior to screening; 2.1 - 3 mSv (inclusive) in the period of 3 years prior to screening, etc. (add 1 year per 1 mSv)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
For Part 1: Absolute bioavailability (F) as percent F (%F) after oral administration as oral to IV ratio of AUC/D (Area under the concentration curve per dose) | Day 1 of Part 1 pre-dose and at multiple time points (up to 3 days) post-dose
For Part 1: AUC of BAY2927088 and [14C]-BAY2927088 | Day 1 of Part 1 pre-dose and at multiple time points (up to 3 days) post-dose
For Part 1: AUC/D of BAY2927088 and [14C]-BAY2927088 | Day 1 of Part 1 pre-dose and at multiple time points (up to 3 days) post-dose
For Part 1: Cmax (maximum concentration) of BAY2927088 and [14C]-BAY2927088 | Day 1 of Part 1 pre-dose and at multiple time points (up to 3 days) post-dose
For Part 1: Cmax/D of BAY2927088 and [14C]-BAY2927088 | Day 1 of Part 1 pre-dose and at multiple time points (up to 3 days) post-dose
For Part 2: Amount of BAY2927088 and its metabolites excreted in urine (%AEur), in feces (%AEfec), and in vomit as a percent of the dose (%AEvom, if applicable) | Day 1 of Part 2 pre-dose and at multiple time points (minimum up to 6 days, maximum up to 6 weeks) post-dose
  Based on radioactivity excreted in urine and feces, and vomit as a percentage of the dose to assess mass balance of total radioactivity
For Part 2: AUC of total radioactivity in plasma and whole blood. (AUC(0-tlast) will be used as primary parameter if mean AUC(tlast-∞) >20% of AUC) | Day 1 of Part 2 pre-dose and at multiple time points (minimum up to 6 days, maximum up to 6 weeks) post-dose
For Part 2: Cmax of total radioactivity in plasma and whole blood | Day 1 of Part 2 pre-dose and at multiple time points (minimum up to 6 days, maximum up to 6 weeks) post-dose
For Part 2: AUC of BAY2927088 in plasma. (AUC[0-tlast] will be used as primary parameter if mean AUC[tlast-∞] >20% of AUC) | Day 1 of Part 2 pre-dose and at multiple time points (minimum up to 6 days, maximum up to 6 weeks) post-dose
For Part 2: Cmax of BAY2927088 in plasma | Day 1 of Part 2 pre-dose and at multiple time points (minimum up to 6 days, maximum up to 6 weeks) post-dose

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAE) and severity of treatment-emergent adverse events | From dosing up to 15 days after last dosing

CONTACTS AND LOCATIONS:
Locations (1):
- ICON plc, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22249